CLINICAL TRIAL: NCT06728683
Title: Assist MH Digital Technologies to Support School Mental Health Care
Acronym: ASSIST-MH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3-C Institute for Social Development (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASSIST MH PI; 1R43MH138260-01 (NIH)
Record Dates: First submitted 2024-11-22; First posted 2024-12-11 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Mental Health Strategies; School Mental Health Services; Digital Technologies; Technology Development

STUDY DESIGN:
Intervention Model Description: Participants in the focus group will all be given the same set of study tasks. They will participate in a 60-minute virtual focus group and then rate the proposed Assist-MH product components. Participants in the pilot test will complete the same study tasks as others in their respective group: one group for providers and one group for students. All providers will (a) attend a brief webinar to review research methods and be trained to use Assist-MH, (b) use Assist-MH for at least 2 weeks with at least 3 students, (c) obtain parent consent for students to use Assist-MH as part of their regular school services, (d) complete pre & post provider outcomes measures, and (e) rate their experiences with the prototype. All students will (a) use Assist-MH, (b) rate their experiences with the prototype via the provider survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASSIST-MH (Experimental): Participants in the pilot test will complete the same study tasks as others in their respective group: one group for providers and one group for students. All providers will (a) attend a brief webinar to review research methods and be trained to use Assist-MH, (b) use Assist-MH for at least 2 weeks with at least 3 students, (c) obtain parent consent for students to use Assist-MH as part of their regular school services, (d) complete pre & post provider outcomes measures, and (e) rate their experiences with the prototype. All students will (a) use Assist-MH, (b) rate their experiences with the prototype via a provider survey.
  Interventions: Other: ASSIST-MH

INTERVENTIONS:
Other: ASSIST-MH — The goal of this SBIR is to create Assist-MH, a new interactive digital support system for SMH providers. Assist-MH will offer an innovative suite of diverse MH strategies to help providers address the clinical needs of youth in distress. In Phase I, the focus will be on tools to address depression and anxiety for students ages 12 to 17 years. These MH problems are among the most common for youth, and have shown increasing prevalence in recent years among this age group. Investigators will conduct user-centered testing to determine the set of MH strategies most needed by SMH providers, create a sampling of these resources, and test the usability and promise of the proposed Assist-MH product prior to Phase II full development and pilot testing.

SUMMARY:
The goal of this SBIR is to develop and test Assist-MH, a new interactive digital support system for SMH providers. Assist-MH will offer SMH treatment resources to help providers implement a more customized treatment plan specific to the student's needs. Based on student areas of need, the system will deliver both provider-led MH strategies to optimize time spent with the student and self-paced digital strategies (video, game-based, interactive) for students to augment in-person treatment and provide unique between-session learning and practice.

DETAILED DESCRIPTION:
This 12-month Phase I project will accomplish three specific objectives: (1) conduct iterative testing with SMH providers, (2) create the fully functioning Assist-MH software prototype, and (3) pilot test the prototype with SMH providers (and their students). The first aim is to gather input from key stakeholders. From those who volunteer, investigators will randomly select 36 participants: 12 providers, 12 supervisors, and 12 administrators. To support diversity and generalizability of initial stakeholder feedback, investigators will stratify random selection to obtain equal participation by gender and 50% non-White participation which is expected to approximate 26% Black, 13% Asian American, and 11% multi-racial or other minority subgroup, with 12% of reporting Latinx/Hispanic ethnicity. Following random selection and consenting, stakeholders will participate in a 60-minute virtual focus group (separately by stakeholder type, 6-8 per group). In a semi-structured fashion, the PI will present initial design concepts and examples for each product component. Focus group discussions will be designed to identify pain points and barriers faced by SMH staff and opportunities to lower barriers to SMH service delivery as well as to gather specific recommendations. Following group participation, stakeholders will rate the value (innovation, usefulness, need), feasibility (time efficient, cost efficient, doable), and acceptability (quality of content, accessibility, scope) of the proposed Assist-MH product components. Ratings will be made on a 5-point scale from 1 (Strongly Disagree) to 5 (Strongly Agree) and mean scores will be calculated across items for each area.

After creating the fully functioning prototype (aim #2), the final aim is to pilot test the prototype with SMH providers serving 12- to 17-year-old students to ensure the product components function as intended and to gather preliminary evidence of the potential value and benefits of the Assist-MH product for supporting SMH service delivery. Using the same recruitment methods described in Aim #1, investigators will nationally recruit and randomly select 40 SMH providers. To participate, providers must provide SMH services to 12- to 17-year-old students. Once accepted into the study, the PI will conduct a brief webinar to review research methods and train providers in Assist-MH. Providers will then use Assist-MH as part of their SMH services for at least 2 weeks with at least 3 students. Providers will be responsible for obtaining parent consent for students to use Assist-MH and evaluate their experience via their provider; no identifying student information will be entered into the system (i.e., tracked by ID). Usage data will be collected by the software to determine prototype use amounts, including time spent for specific tasks and number of times each component is accessed. The system will also collect provider and student interactions with treatment strategies. 3C will also track number and type of technical assistance (TA) requests during the pilot test period (e.g., phone and email requests to technical support staff). The following set of measures will be collected before and after the trial period. Each measure is supported by prior studies showing internal consistency, reliability, and content validity with providers. For provider outcomes, investigators will assess three areas found to be associated with the quality of care among MH providers, and which investigators expect to change as a function of access to Assist-MH: Perceived Quality of Care scale, Self-efficacy (via Comfort and Skills survey), and Emotional Exhaustion subscale of the Human Service Provider version of the Maslach Burnout Inventory. Lastly, providers will rate their experiences with the prototype. Ratings will be made on a 5-pt scale (1=Strongly Disagree to 5=Strongly Agree) to assess each component and the overall prototype in each of the following areas: usability (e.g., user friendly, easy to navigate, engaging), feasibility (e.g., time efficient, doable), and value (e.g., quality, innovation, effectiveness for intended purpose). Providers will also ask students questions to report on their experiences using the prototype. Mean scores will be calculated across items for each area. Open-ended questions will also be included to gather qualitative comments and recommendations.

ELIGIBILITY:
Inclusion Criteria:

* must be a SMH provider (providing services to 12- to 17-year-old students) or a student (12 to 17 years old)
* must have access to internet
* must be English language proficient.
* No one will be excluded based on gender, race, or ethnic background.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Pilot prototype evaluation | Within 1 week of study completion
  Providers will rate their experiences with the prototype. Ratings will be made on a 5-pt scale (1=Strongly Disagree to 5=Strongly Agree) to assess each component and the overall prototype in each of the following areas: usability (e.g., user friendly, easy to navigate, engaging), feasibility (e.g., time efficient, doable), and value (e.g., quality, innovation, effectiveness for intended purpose). The 24 items will be computed into a summary score ranging from 1-5 to reflect mean ratings. A higher rating indicates stronger support for the Assist-MH product. Providers will ask students who participated in reviewing the strategies questions about their experience with the prototype. Providers will fill in their responses on the pilot prototype evaluation.

SECONDARY OUTCOMES:
Perceived Quality of Care scale | 2 months apart, as Pre- and Post-Test
  Will be used to measure providers' self-perception of the level of quality of care they provide to students. Providers rate 22 items on a 6-pt scale (1=Never to 6=Always) related to person-centered care (e.g., helped student meet personal/treatment goal) and discordant care (e.g., delayed response to requests, made mistakes). A mean score will be computed. Perceived quality of care score means range from 1 to 6. Higher mean score reflects higher perceived quality.
Comfort & Skills survey | 2 months apart, as Pre- and Post-Test
  Will be used to assess providers' level of confidence and self-perceived skills with SMH treatment planning and delivery, such as "I know how to judge severity of student MH problems," "I can deliver services that help a student," and "I am confident in my ability to provide evidence-based care." Ratings are made on a 5-pt scale (1=Not true to 5=Very true). A mean score will be computed. Comfort and skill score means range from 1 to 5. Higher score reflects greater self-efficacy.
Emotional Exhaustion subscale | 2 months apart, as Pre- and Post-Test
  Providers will complete the 9-item subscale of the Human Service Provider version of the Maslach Burnout Inventory (MBI-HSS). Providers rate how often they feel each item (e.g., "I feel emotionally drained from my work") on a 7-pt scale (1=Never to 7=Everyday). A mean score will be computed. Emotional Exhaustion score means range from 1 to 7. Higher scores indicate higher emotional exhaustion, a key component of burnout among MH providers.
Provider Reported Student Usability ratings | Within 1 week of study completion
  Students will rate their experiences with the prototype. Ratings will be made on a 5-pt scale (1=Strongly Disagree to 5=Strongly Agree) to assess the usability of the Assist-MH prototype. The 4 items will be computed into a summary score ranging from 1-5 to reflect mean ratings. A higher rating indicates stronger support for the Assist-MH product.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa E DeRosier, PhD, Principal Investigator — 3-C Institute for Social Development
Locations (1):
- 3-C Institute for Social Development, Inc, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided